CLINICAL TRIAL: NCT03315806
Title: Effect of Beetroot Juice Consumption on Endothelial Function and Tissue Oxygen Saturation in Pregnant
Brief Title: Pregnancy, Nitrate, Endothelial Function and Tissue Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, PhD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 56732216.5.0000.5699
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy
Keywords: Dietary nitrate; Nitrate; Flow-mediated dilation; Tissue oxygen saturation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot Juice (Active Comparator): Beetroot juice containing 9 mmol of nitrate per dose
  Interventions: Other: Beetroot juice
- Placebo juice (nitrate depleted) (Placebo Comparator): Beetroot juice nitrate-depleted
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Beetroot juice — 140 mL of beetroot juice cointaning approximately 9 mmol of nitrate
  Arms: Beetroot Juice
Other: Placebo — 140 mL of beetroot juice isent of nitrate
  Arms: Placebo juice (nitrate depleted)

SUMMARY:
Adequate macro and microvascular endothelial function during pregnancy is essential for the normal placental development and growing fetus. Beetroot juice (BJ) promotes improvement ins this parameters in no-pregnant individuals, however the beneficial effect did not avaliated in pregnant. The present study evaluated effects of BJ on macro and microvascular endothelial function in pregnant. Twelve pregnant were submitted to BJ and nitrate-depleted juice (PLA) interventions. Brachial flow-mediated dilation (FMD) and muscle oxygenation were measured 120 min after interventions. Urinary nitrate, nitrite were measured at baseline and 120 min after interventions.

ELIGIBILITY:
Inclusion Criteria:

* gestation between 20 and 35 weeks;
* over 18 years

Exclusion Criteria:

* diabetes mellitus and gestational diabetes;
* hypertensive syndromes;
* HIV positive;
* liver or kidney disease;
* beetroot allergy;
* use of antioxidants and medicament that alter endothelial function;
* use of antibiotics up to 2 weeks before the visits and using.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Macro endothelial function | Evaluated 120 minutes after the nutritional intervention
  Flow-mediated dilation (FMD)
Micro endothelial function | Evaluated 140 minutes after the nutritional intervention
  Tissue oxygen saturation parameters
Nitrate urinary | Evaluated 150 minutes after the nutritional intervention